CLINICAL TRIAL: NCT00563615
Title: Study of Effect of Tegaserod on Small and Large Bowel Transit by Scintigraphic Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KW/FR/03-030; HARECCTR0500026
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Constipation
Keywords: Constipation (idiopathic)
MeSH Terms: conditions — Constipation | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Functional constipation is a common problem in Hong Kong. In a recent telephone survey, the prevalence of constipation as defined by Rome II criteria was 14%. Apart from organic, metabolic, neurological and drug induced causes, constipation most often arises from 2 disorders of colorectal motility: slow transit constipation or pelvic floor dysfunction or both. In the position statement from the American Gastroenterological Association , colon transit study was recommended to differentiate slow transit constipation from pelvic floor dysfunction. The management algorithm for normal transit and slow transit constipation was different and surgery should be considered for patients with slow transit constipation. In a recent paper by Bonapace , scintigraphy could be used to study both gastric, small bowel and large bowel transit time. The clinical diagnosis was changed in 51% of cases of constipation after scintigraphy and patient management such as adding a prokinetic agent, referral to biofeedback center, decision on surgery was affected in 64% of cases.

Tegaserod is a recently approved prokinetic agent to be marketed in Hong Kong for the management of patients with constipation predominant irritable bowel syndrome (C-IBS). In a paper from Mayo clinic based on scintigraphic examination, tegaserod 2mg bd accelerates orocaecal transit in C-IBS patients. However studies in functional constipation basing on tegaserod 6 mg twice daily has not been published yet. Therefore, the Gastroenterology team and nuclear medicine teams of Princess Margaret Hospital, Gastroenterology teams of Caritas Medical Center and Yan Chai Hospital decide to study small and large bowel transit in functional constipation patients by scintigraphy. The efficacy of tegaserod in improving bowel transit is also examined in this randomized double blind placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* History of functional constipation as proposed by the Rome II Criteria and the usual frequency of spontaneous bowel motion must be equal or less than 2 times /week.
* An endoscopic/radiologic bowel evaluation (colonoscopic examination and/or a sigmoidoscopy + barium enema) is required in patients older than 40 years. This evaluation must have been performed within the past 5 years. In addition, there should not be history or evidence of weight loss, anemia or rectal bleeding since the evaluation was performed.

Note: For patients who require these procedures, these tests should be performed after the patient has signed informed consent and at least 7 days PRIOR to the start of the diaries (washout period). The 7-day window is to allow the patient to recuperate prior to collecting baseline data.

A copy of the report should be placed in the patient source document.

* Patients who are able to communicate well with the investigator and to comply with the requirements for the entire study, including the withdrawal period.
* Patients who provide written informed consent before participating in the study after being given a full description of the study.

Exclusion Criteria:

* Medications known to affect gastrointestinal transit before 1 week of the treatment phase of the study.
* With clinical evidence (including physical exam, vital signs, ECG, laboratory tests) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematology, endocrine or metabolic disorders, neurologic disease, or of any disease that may interfere with the patient successfully completing the study.
* Existence of surgical or medical conditions which interfere with the absorption, distribution, metabolism and excretion of the study medication.
* With hypo or hyper thyroidism (clinically significant abnormal TSH level at screening).
* With symptoms of a significant clinical illness in the two weeks preceding baseline.
* With other relevant intercurrent medical condition that may interfere with the objectives of the study.
* Women who are pregnant or breast-feeding.
* With evidence or history of drug or alcohol abuse within the past 12 months.
* Who received another investigational drug within the 30 days prior to entry in the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-11; Study Completion 2006-10 (Estimated)

PRIMARY OUTCOMES:
Small and large bowel transit time | 2 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ambrose CP Kwan, Dr, Principal Investigator — Department of Medicine and Geriatrics, Unit A, Princess Margaret Hospital
Locations (3):
- China (3):
  - Caritas Medical Centre, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Yan Chai Hospital, Hong Kong